CLINICAL TRIAL: NCT00703625
Title: Phase I Study of Docetaxel and Temsirolimus in Resistant Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0444
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Resistant Solid Malignancies
MeSH Terms: interventions — temsirolimus; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Temsirolimus IV 15 mg weekly
  Docetaxel 60 mg/m2 IV once every three weeks.
  Interventions: Drug: Temsirolimus; Drug: Docetaxel
- Cohort 2 (Experimental): Temsirolimus IV 25 mg weekly
  Docetaxel IV 60 mg/m2 once every 3 weeks
  Interventions: Drug: Temsirolimus; Drug: Docetaxel
- Cohort 1A (Experimental): Temsirolimus IV 15 mg weekly
  Docetaxel IV 50 mg/m2 every 3 weeks.
  Interventions: Drug: Temsirolimus; Drug: Docetaxel

INTERVENTIONS:
Drug: Temsirolimus
  Other Names: Torisel; CCI-779
Drug: Docetaxel
  Other Names: Taxotere

SUMMARY:
Rationale:

The Mammalian Target of Rapamycin (mTOR) is a large polypeptide serine/threonine kinase of 289 kDa; kinases have been shown to be important regulators of cancer cell cycle, proliferation, invasion, and angiogenesis, and mTOR has been shown to have a key role in the signaling of malignant cell growth, proliferation, differentiation, migration, and survival. Inhibition of mTOR would result in arrest of cell growth in the G1 phase of the cell cycle.

Temsirolimus (CCI-779) is a soluble ester analogue of rapamycin (sirolimus) which has shown impressive in vitro and in vivo cytostatic activity in selectively inhibiting mTOR. In animal models, temsirolimus has demonstrated an impressive cytostatic effect on a wide variety of cancer cells. In vitro, it inhibited the growth of human T-cell leukemia, glioblastoma, melanoma, prostate, breast, renal cell, and pancreatic cells, all of which showed particular sensitivity to temsirolimus, with significant growth inhibition at concentrations of less that 0.01micrometers. In Phase I trials, temsirolimus has been investigated as a single agent on a weekly schedule as well as daily for 5 days every other week, and evidence of activity was observed over the entire dose range (15 - 220 mg/m2) in patients with both breast and renal cancer. There was no apparent relationship between exposure and clinical benefit, suggesting that the inhibition of mTOR may be achieved at doses well below dose levels that result in dose limiting toxicities. Major tumor responses were noted in Phase I trials in patients previously treated with lung, breast, renal as well as neuroendocrine tumors. Minor responses were noted in soft tissue sarcoma, endometrial, and cervical carcinoma.

Docetaxel is a taxane analog which is active against many solid tumors including breast, non-small cell lung, prostate, gastric, ovarian, head and neck, and pancreatic cancers, soft tissue sarcoma, and melanoma. It has been shown in several Phase III studies to have clinically significant activity in several solid tumors.

We propose treating patients with resistant solid malignancies with docetaxel and temsirolimus. In a study using human breast cancer cell lines, mTOR inhibition with rapamycin had a synergistic cytotoxic effect with paclitaxel. Given the novel mechanism of action of mTOR inhibitors and known synergistic activity of an mTOR inhibitor, rapamycin, with a taxane, paclitaxel, in vitro, we envision that this regimen would be highly active in patients with solid tumor malignancies.

Objectives:

Primary

* To define the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies.
* To determine the incidence and severity of other toxicities of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies.

Secondary

* To assess the pharmacokinetic profile of temsirolimus in combination with pegylated liposomal doxorubicin.
* To determine any anti-tumor activity and response to the combination of temsirolimus and pegylated liposomal doxorubicin in treatment of patients with resistant solid malignancies.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

* Patients must have a histologically or cytologically proven solid malignancy which is resistant to conventional therapy or for which no effective therapy is known.
* Patients with measurable or non-measurable disease are eligible for entry to this study. In addition, patients without measurable or non-measurable disease are also eligible.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. Neuropathy must have recovered to grade 1. No chemotherapy or radiotherapy may be given within 4 weeks prior to the start of protocol treatment.
* Patients must be ≥18 years old.
* ECOG 0-2 at study entry.
* Patients must have a life expectancy of greater than 8 weeks.
* Required Laboratory Values:
* absolute neutrophil count ≥1,500/mm3
* platelets ≥100,000/mm3
* hemoglobin ≥9.0 g/dL
* total bilirubin ≤1.5 x ULN
* AST(SGOT)/ALT(SGPT) ≤1.5 x ULN (≤2.5 x ULN for patients with liver metastases
* alkaline phosphatase ≤2.5 x ULN
* creatinine ≤1.5 x ULN OR
* creatinine clearance ≥60 mL/min/1.732 for patients with creatinine levels above 2.0 mg/dl
* serum cholesterol ≤350 mg/dL /9.0 mmol/L (fasting)
* triglycerides ≤400 mg/dL (fasting)*
* albumin ≥3.0 mg/dL
* PT/INR ≤1.5, unless the patient is on full dose warfarin or stable dose of LMW heparin with a therapeutic INR of >1.5 - ≤3
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels.
* Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin) are not eligible for this trial.
* For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women are not eligible.
* Patients must not have active CNS disease.
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Patients must have signed a Washington University, Human Research Protection Office (HRPO) approved informed consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03-08 (Actual); Primary Completion 2011-05-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies. | After completion of cycle 1 by all patients
To determine the incidence and severity of other toxicities of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies. | 30 days after completion of treatment

SECONDARY OUTCOMES:
To assess the pharmacokinetic profile of temsirolimus in combination with pegylated liposomal doxorubicin. | Through cycle 2 day 8
  cycle 1 day 1, cycle 2 day 1 (pre-dose, 0.5 hours before end of temsirolimus infusion, 1.5 hours after start of temsirolimus infusion, 5 hours after start of temsirolimus infusion), cycle 2 day 3, cycle 2 day 5, and cycle 2 day 8
To determine any anti-tumor activity and response to the combination of temsirolimus and pegylated liposomal doxorubicin in treatment of patients with resistant solid malignancies. | End of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Wullschleger S, Loewith R, Hall MN. TOR signaling in growth and metabolism. Cell. 2006 Feb 10;124(3):471-84. doi: 10.1016/j.cell.2006.01.016. PMID 16469695
- [Background] Adjei AA, Hidalgo M. Intracellular signal transduction pathway proteins as targets for cancer therapy. J Clin Oncol. 2005 Aug 10;23(23):5386-403. doi: 10.1200/JCO.2005.23.648. Epub 2005 Jun 27. PMID 15983388
- [Background] Smolewski P. Recent developments in targeting the mammalian target of rapamycin (mTOR) kinase pathway. Anticancer Drugs. 2006 Jun;17(5):487-94. doi: 10.1097/00001813-200606000-00001. PMID 16702804
- [Background] Thomas GV. mTOR and cancer: reason for dancing at the crossroads? Curr Opin Genet Dev. 2006 Feb;16(1):78-84. doi: 10.1016/j.gde.2005.12.003. Epub 2005 Dec 15. PMID 16359855
- [Background] Elit L. CCI-779 Wyeth. Curr Opin Investig Drugs. 2002 Aug;3(8):1249-53. PMID 12211424
- [Background] Huang S, Houghton PJ. Targeting mTOR signaling for cancer therapy. Curr Opin Pharmacol. 2003 Aug;3(4):371-7. doi: 10.1016/s1471-4892(03)00071-7. PMID 12901945
- [Background] Sawyers CL. Will mTOR inhibitors make it as cancer drugs? Cancer Cell. 2003 Nov;4(5):343-8. doi: 10.1016/s1535-6108(03)00275-7. No abstract available. PMID 14667501
- [Background] Del Bufalo D, Ciuffreda L, Trisciuoglio D, Desideri M, Cognetti F, Zupi G, Milella M. Antiangiogenic potential of the Mammalian target of rapamycin inhibitor temsirolimus. Cancer Res. 2006 Jun 1;66(11):5549-54. doi: 10.1158/0008-5472.CAN-05-2825. PMID 16740688
- [Background] Chan S. Targeting the mammalian target of rapamycin (mTOR): a new approach to treating cancer. Br J Cancer. 2004 Oct 18;91(8):1420-4. doi: 10.1038/sj.bjc.6602162. PMID 15365568
- [Background] Teachey DT, Obzut DA, Cooperman J, Fang J, Carroll M, Choi JK, Houghton PJ, Brown VI, Grupp SA. The mTOR inhibitor CCI-779 induces apoptosis and inhibits growth in preclinical models of primary adult human ALL. Blood. 2006 Feb 1;107(3):1149-55. doi: 10.1182/blood-2005-05-1935. Epub 2005 Sep 29. PMID 16195324
- [Background] Hidalgo M, Rowinsky E, Erlichmann C, et al. A Phase I and Pharmacological Study of CCI-779, a Rapamycin Ester Cell Cycle Inhibitor. Annals of Oncology 11(Suppl4): 133, 2000.
- [Background] Raymond E, Alexandre J, Faivre S, Vera K, Materman E, Boni J, Leister C, Korth-Bradley J, Hanauske A, Armand JP. Safety and pharmacokinetics of escalated doses of weekly intravenous infusion of CCI-779, a novel mTOR inhibitor, in patients with cancer. J Clin Oncol. 2004 Jun 15;22(12):2336-47. doi: 10.1200/JCO.2004.08.116. Epub 2004 May 10. PMID 15136596
- [Background] Punt CJ, Boni J, Bruntsch U, Peters M, Thielert C. Phase I and pharmacokinetic study of CCI-779, a novel cytostatic cell-cycle inhibitor, in combination with 5-fluorouracil and leucovorin in patients with advanced solid tumors. Ann Oncol. 2003 Jun;14(6):931-7. doi: 10.1093/annonc/mdg248. PMID 12796032
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Oza A, Elit L, Biagi J, Gotlieb W, Tonkin K, Tsao MN, et al. A Phase II Study of Temsirolimus (CCI-779) in Patients with Metastatic and/or Recurrent Endometrial Cancer. Clinical Cancer Research 11: 9099s, 2005
- [Background] Chan S, Scheulen ME, Johnston S, Mross K, Cardoso F, Dittrich C, Eiermann W, Hess D, Morant R, Semiglazov V, Borner M, Salzberg M, Ostapenko V, Illiger HJ, Behringer D, Bardy-Bouxin N, Boni J, Kong S, Cincotta M, Moore L. Phase II study of temsirolimus (CCI-779), a novel inhibitor of mTOR, in heavily pretreated patients with locally advanced or metastatic breast cancer. J Clin Oncol. 2005 Aug 10;23(23):5314-22. doi: 10.1200/JCO.2005.66.130. Epub 2005 Jun 13. PMID 15955899
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Pandya KJ, Levy DE, Hidalgo M, et al. A Randomized, Phase II ECOG Trial of Two Dose Levels of Temsirolimus (CCI-779) in Patients with Extensive Stage Small Cell Lung Cancer in Remission After Induction Chemotherapy. A Preliminary Report. Journal of Clinical Oncology. ASCO Annual Meeting Proceedings; 23: 7005, 2005.
- [Background] Margolin K, Longmate J, Baratta T, Synold T, Christensen S, Weber J, Gajewski T, Quirt I, Doroshow JH. CCI-779 in metastatic melanoma: a phase II trial of the California Cancer Consortium. Cancer. 2005 Sep 1;104(5):1045-8. doi: 10.1002/cncr.21265. PMID 16007689
- [Background] Chang SM, Wen P, Cloughesy T, Greenberg H, Schiff D, Conrad C, Fink K, Robins HI, De Angelis L, Raizer J, Hess K, Aldape K, Lamborn KR, Kuhn J, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Phase II study of CCI-779 in patients with recurrent glioblastoma multiforme. Invest New Drugs. 2005 Aug;23(4):357-61. doi: 10.1007/s10637-005-1444-0. PMID 16012795
- [Background] Hudes G, Carducci M, Tomczak P, et al. A Phase 3, Randomized, 3-arm Study of Temsirolimus (TEMSR) or Interferon-alpha (IFN) or the Combination of TEMSR + IFN in the Treatment of First-Line, Poor-Risk Patients with Advanced Renal Cell Carcinoma (adv RCC). Journal of Clinical Oncology, ASCO Annual Meeting Proceedings; 24: LBA4, 2006.
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Ramaswamy B, Puhalla S. Docetaxel: a tubulin-stabilizing agent approved for the management of several solid tumors. Drugs Today (Barc). 2006 Apr;42(4):265-79. doi: 10.1358/dot.2006.42.4.968648. PMID 16703123
- [Background] Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F, Kalman L, Miller V, Lee JS, Moore M, Gandara D, Karp D, Vokes E, Kris M, Kim Y, Gamza F, Hammershaimb L. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol. 2000 Jun;18(12):2354-62. doi: 10.1200/JCO.2000.18.12.2354. PMID 10856094
- [Background] Jones SE, Erban J, Overmoyer B, Budd GT, Hutchins L, Lower E, Laufman L, Sundaram S, Urba WJ, Pritchard KI, Mennel R, Richards D, Olsen S, Meyers ML, Ravdin PM. Randomized phase III study of docetaxel compared with paclitaxel in metastatic breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5542-51. doi: 10.1200/JCO.2005.02.027. PMID 16110015
- [Background] Charles KA, Rivory LP, Stockler MR, Beale P, Beith J, Boyer M, Clarke SJ. Predicting the toxicity of weekly docetaxel in advanced cancer. Clin Pharmacokinet. 2006;45(6):611-22. doi: 10.2165/00003088-200645060-00004. PMID 16719542
- [Background] Chen YM, Shih JF, Perng RP, Tsai CM, Whang-Peng J. A randomized trial of different docetaxel schedules in non-small cell lung cancer patients who failed previous platinum-based chemotherapy. Chest. 2006 Apr;129(4):1031-8. doi: 10.1378/chest.129.4.1031. PMID 16608954
- [Background] Schuette W, Nagel S, Blankenburg T, Lautenschlaeger C, Hans K, Schmidt EW, Dittrich I, Schweisfurth H, von Weikersthal LF, Raghavachar A, Reissig A, Serke M. Phase III study of second-line chemotherapy for advanced non-small-cell lung cancer with weekly compared with 3-weekly docetaxel. J Clin Oncol. 2005 Nov 20;23(33):8389-95. doi: 10.1200/JCO.2005.02.3739. PMID 16293869
- [Background] Ford HE, Yap YS, Miles DW, Makris A, Hall M, Miller L, Harries M, Smith IE, Johnston SR. A phase II study of weekly docetaxel in patients with anthracycline pretreated metastatic breast cancer. Cancer Chemother Pharmacol. 2006 Dec;58(6):809-15. doi: 10.1007/s00280-006-0222-9. Epub 2006 Mar 10. PMID 16528527
- [Background] Mondesire WH, Jian W, Zhang H, Ensor J, Hung MC, Mills GB, Meric-Bernstam F. Targeting mammalian target of rapamycin synergistically enhances chemotherapy-induced cytotoxicity in breast cancer cells. Clin Cancer Res. 2004 Oct 15;10(20):7031-42. doi: 10.1158/1078-0432.CCR-04-0361. PMID 15501983
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Yazbeck VY, Georgakis GV, Li Y, and Younes A. The mTOR Inhibitor CCI-779 (Temsirolimus) Downregulates p21 and Induces Cell Cycle Arrest and Autophagy in Mantle Cell Lymphoma (MCL). Journal of Clinical Oncology, ASCO Annual Meeting Proceedings; 24:7573, 2006.
- [Background] Duran I, Siu LL, Oza AM, Chung TB, Sturgeon J, Townsley CA, Pond GR, Seymour L, Niroumand M. Characterisation of the lung toxicity of the cell cycle inhibitor temsirolimus. Eur J Cancer. 2006 Aug;42(12):1875-80. doi: 10.1016/j.ejca.2006.03.015. Epub 2006 Jun 27. PMID 16806903
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu